CLINICAL TRIAL: NCT00719095
Title: Effective Treatment for Prescription Opioid Abuse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Stacey C. Sigmon, Ph.D., University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01DA019989 (NIH); R01DA019989 (NIH)
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2008-07

CONDITIONS: Prescription Opioid Dependence
Keywords: prescription opioid; opioid detoxification; buprenorphine; naltrexone; community reinforcement approach; prescription opioid abuse
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1-week buprenorphine taper (Experimental): 1-week buprenorphine taper + behavioral therapy + urine toxicology
  Interventions: Drug: buprenorphine taper followed by naltrexone maintenance; Behavioral: Behavioral therapy
- 2-week buprenorphine taper (Experimental): 2-week buprenorphine taper + behavioral therapy + urine toxicology
  Interventions: Drug: buprenorphine taper followed by naltrexone maintenance; Behavioral: Behavioral therapy
- 4-week buprenorphine taper (Experimental): 4-week buprenorphine taper + behavioral therapy + urine toxicology
  Interventions: Drug: buprenorphine taper followed by naltrexone maintenance; Behavioral: Behavioral therapy

INTERVENTIONS:
Drug: buprenorphine taper followed by naltrexone maintenance — direct comparison of 1-, 2- and 4-week durations of buprenorphine taper for treating prescription opioid abusers; those who successfully taper without resumption of illicit opioid use are subsequently transitioned to oral naltrexone therapy for the remainder of the 12-week trial; all participants receive a platform of intensive individual behavioral therapy and on-site urinalysis monitoring throughout the trial
Behavioral: Behavioral therapy

SUMMARY:
There has been an alarming increase in abuse of prescription opioids in recent years. This project aims to develop an effective outpatient treatment for prescription opioid (PO) abuse that combines an intensive behavioral therapy with a pharmacotherapy regimen of buprenorphine detoxification and naltrexone maintenance.

DETAILED DESCRIPTION:
There has been an alarming increase in abuse of prescription opioids in recent years. This project aims to develop an effective outpatient treatment for prescription opioid (PO) abuse that combines an intensive behavioral therapy with a pharmacotherapy regimen of buprenorphine detoxification and naltrexone maintenance. Aim 1) Conduct a randomized, three-parallel-groups clinical trial (Study 1) to determine a buprenorphine dose-tapering schedule that prevents the poor retention and relapse that undermine many opioid detoxification regimens. Aim 2) Conduct a randomized, three-parallel-groups clinical trial (Study 2) to determine a duration of naltrexone therapy that sustains opioid abstinence following the buprenorphine detoxification.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion in the proposed studies, subjects must be > 18 years old and in good health. Subjects must meet DSM-IV criteria for opioid dependence and FDA qualification criteria for buprenorphine treatment, including a history of opioid dependence and significant current opioid use (i.e., opioid-positive urines). Subjects must also be seeking or willing to accept opioid detoxification.

Exclusion Criteria:

* Because the primary focus of the proposed research is to develop an efficacious intervention for prescription opioid abuse that employs a buprenorphine taper and subsequent naltrexone maintenance, individuals who require ongoing opioid therapy for pain or other chronic medical conditions will be excluded from participating.
* Individuals with evidence of an active psychiatric disorder that may interfere with consent or participation in the research (e.g., psychosis, manic-depressive illness, organic psychiatric disorders), significant medical illness (e.g., cardiovascular disease) or who are pregnant or nursing will be excluded from participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2006-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
percentage of subjects abstinent from all opioids through the final day of detoxification | up to 12-week trial

SECONDARY OUTCOMES:
percentage of subjects retained in treatment through the final day of detoxification | up to 12-week trial

CONTACTS AND LOCATIONS:
Overall Officials: Stacey C. Sigmon, Ph.D., Principal Investigator — University of Vermont, Department of Psychiatry
Locations (1):
- Substance Abuse Treatment Center, University of Vermont, Burlington, Vermont, United States

REFERENCES:
- [Derived] Sigmon SC, Dunn KE, Saulsgiver K, Patrick ME, Badger GJ, Heil SH, Brooklyn JR, Higgins ST. A randomized, double-blind evaluation of buprenorphine taper duration in primary prescription opioid abusers. JAMA Psychiatry. 2013 Dec;70(12):1347-54. doi: 10.1001/jamapsychiatry.2013.2216. PMID 24153411